CLINICAL TRIAL: NCT02703415
Title: Comparison Of Immune Response And Analgesic Effects Of Caudally Administrated Tramadol In Pediatric Lower Abdominal Surgery
Brief Title: Immune Response of Caudally Administrated Tramadol In Pediatric Lower Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB000087400
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Acute Pain
Keywords: immune; interleukin; tramadol; postoperartive analgesia; pediatric; caudal bupivacaine
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Tramadol; tamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Active Comparator): caudal Bupivacaine
  Interventions: Drug: Bupivacaine
- Tramadol (Active Comparator): caudal Tramadol
  Interventions: Drug: Bupivacaine; Drug: Tramadol

INTERVENTIONS:
Drug: Bupivacaine — caudal block with bupivacaine (0.25%) 1mg/kg
  Other Names: Marcaine
Drug: Tramadol — caudal block with tramadol 1 mg/kg
  Other Names: Tamol
  Arms: Tramadol

SUMMARY:
Management of acute pain is one of the most important tasks of perioperative pediatric anesthesia. The alleviation of pain has been defined by the Society of Pediatric Anesthesia, on its 15th annual meeting as a basic human right, irrespective of age, treatment primary service responsible for the patient care. Pro-inflammatory cytokines increased by surgical trauma indirectly modulate pain through the release of substances like nitric oxide, oxygen free radicals, prostaglandins, and excitatory amino acids, inducing peripheral and central sensitivity and hyperalgesia. There has been growing interest in determining the possible immune consequences of analgesic administration for the management of postoperative pain

DETAILED DESCRIPTION:
60 children aged 3-10 years undergoing lower abdominal surgery will be randomized into 2 groups (30 patients in each group) to receive caudal block with bupivacaine (0.25%) 1mg/kg (group 1) plus tramadol 1mg/kg (group 2) just after the induction of general anesthesia without premedication. All children will be assessed for the post operative immune response by measuring interleukin 6 and 10 (IL-6 and IL-10) and Tumour Necrosing Factor-α (TNF-α) using enzyme-linked immunosorbent assay (ELISA) technique one hour preoperatively and three hours after incision.

ELIGIBILITY:
Inclusion Criteria:

lower abdominal operation

Exclusion Criteria:

Any systemic disease that might compromise the immune system severe coagulation disorder true allergy to local anesthetics patients with major malformations of the lower spine or meninges any cutaneous or subcutaneous lesion at the site of injection unplanned reoperation, or reoperation within three months Diabetes Melliutes

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
post operative immune response | within the first three days postoperatiely
  post operative immune response by measuring interleukin 6 (IL-6) using enzyme-linked immunosorbent assay (ELISA) technique, serum cortisol, C-reactive protein (CRP), and phopholipase A2 (PLA2) one hour preoperatively, end of anesthesia, 1st post- operative day, and 3rd post- operative day

SECONDARY OUTCOMES:
. Post operative pain intensity | within the first postoperative day
  Post operative pain intensity with the FLACC pain scale for five categories (F) Face, (L) Legs, (A) Activity, (C) Cry, (C) consolability will be assessed.
Time of first supplemental analgesia | within the first postoperative day
  Time of first supplemental analgesia
sedation score | Within the first 24 hours
  Sedation assessment after extubation by Richmond Agitation Sedation Scale (RASS)
side effects | Within the first 24 hours
  hypotension, vomiting, pruritus, urinary retention or motor weakness will be recorded.
Leucocyte count | within the first three days postoperatiely
  Leucocyte count and the percentages of neutrophils, lymphocytes and monocytes at one hour preoperatively, end of anesthesia, 1st post- operative day, and 3rd post- operative day

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided